CLINICAL TRIAL: NCT05209841
Title: Heparinization vs Salinization of the Peripheral Venous Catheter: a Randomized Clinical Trial
Brief Title: Heparinization vs Salinization of the Peripheral Venous Catheter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CSAPG-18
Record Dates: First submitted 2021-12-29; First posted 2022-01-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Catheter Complications
Keywords: Catheterization, Peripheral; Catheter Obstruction
MeSH Terms: interventions — Heparin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter sealing with low dose heparin (Experimental): Catheters will be sealed with 3mL of Fibrillin Ⓡ (heparin 20UI/mL)
  Interventions: Drug: Low dose heparin
- Catheter sealing with normal saline (Active Comparator): Catheters will be sealed with 3mL of 0.9% sodium chloride
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Low dose heparin — Catheters will be sealed with 3 mL of Fibrillin Ⓡ (heparin 20UI/mL)
  Arms: Catheter sealing with low dose heparin
Drug: Normal saline — Catheters will be sealed with 3mL of 0.9% sodium chloride
  Arms: Catheter sealing with normal saline

SUMMARY:
Randomized, double-blind clinical trial to compare the efficacy of catheter sealing with saline, compared to low-dose heparin. 3,450 patients hospitalized at the Hospital Residencia Sant Camil, in Catalonia (Spain), will be randomized to each branch of study. The primary outcome will be the percentage of catheters removed due to obstruction in each branch of study. As secondary outcomes, the number of catheter-associated phlebitis, catheter-associated bacetrihemia, extravasation, and catheter loss will be measured. For the primary outcome, a superiority analysis will be carried out in terms of the percentage of obstructed catheters in each branch of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 yo, admitted to the Hospital Residencia Sant Camil
* Patients with at least one peripheral venous line for discontinuous treatment, which has not been channeled in a medical emergency situation.
* Written informed consent

Exclusion Criteria:

* Allergy to heparin
* Patients treated with unfractionated sodium heparin.
* Patients in dialysis
* Patients with a venous catheter indicated for diagnosis tests.
* Patients with a venous catheter indicated for blood transfusion
* Severe heparin-induced thrombocytopenia in recent months
* Active uncontrollable bleeding during admission
* Brain aneurysm or dissecting aorta, except in association with corrective surgery.
* Confirmed / suspected cerebrovascular hemorrhage
* Severe uncontrolled hypertension
* Severe alterations in platelet coagulation <30,000, TP> 1.7 APTT ratio> 1.7 ratio.
* Patient included in another clinical trial with drugs or procedures that may affect the patency of venous catheters.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3450 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of obstructed catheters | From date of randomization through the date of hospital discharge, an average of 10 days.
  percentage of obstructed catheters

SECONDARY OUTCOMES:
Number of catheter-associated phlebitis | From date of randomization through the date of hospital discharge, an average of 10 days.
  Number of catheter-associated phlebitis
Number of catheter-associated bacterihemia episodes | From date of randomization through the date of hospital discharge, an average of 10 days.
  Number of catheter-associated bacterihemia episodes
Number of catheter loss due to extravasation | From date of randomization through the date of hospital discharge, an average of 10 days.
  Number of catheter loss due to extravasation

CONTACTS AND LOCATIONS:
Overall Officials: Esther Moreno Rubio, Principal Investigator — CSAPG
Locations (1):
- Hospital Residència Sant Camil, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research proposels and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.